CLINICAL TRIAL: NCT06850025
Title: Heat Waves, Urban Heat Islands, and Wellbeing and Health: a Mobile Sensing Approach (H3Sensing)
Brief Title: Heat Waves, Urban Heat Islands, and Wellbeing and Health: a Mobile Sensing Approach
Acronym: H3Sensing
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C22-60; 2022-A02108-35 (Other: IDRCB)
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: General Population, no Specific Condition
Keywords: Heat waves; Urban Heat Islands; Wellbeing; Health; Thermoregulation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 180 participants from the Grand Paris area: 180 participants recruited in the Grand Paris area through web and social network advertisements.

SUMMARY:
The first objective of H3Sensing is to investigate outdoor environmental, building, dwelling, situational, and behavioral determinants of objectively assessed personal heat stress over daily movements during warm periods.

The second aim is to investigate how these heat stress determinants and momentary and cumulated heat stress itself are related to physiological indicators of heat stress, sleep, thermal discomfort, and well-being.

DETAILED DESCRIPTION:
While the number of heat wave days in France will likely continue to increase over the century, extreme heat is associated with excess mortality and morbidity in urban heat islands. The first objective of H3Sensing is to investigate outdoor environmental, building, dwelling, situational, and behavioral determinants of objectively assessed personal heat stress over daily movements during warm periods. We will explore environmental determinants associated with micro-urban heat islands at an unprecedented level of accuracy; we will assess building and dwelling characteristics associated with in-home heat stress; and we will examine how daily activities (trips, etc.) and practices (how people dress, manage heat at home) contribute to heat stress. The second aim is to investigate how these heat stress determinants and momentary and cumulated heat stress itself are related to physiological indicators of heat stress, sleep, thermal discomfort, and well-being. One hundred eighty (180) participants recruited through internet advertisements will be followed over 4 day periods in March-May and then a second time in June-September 2025. Research assistants will use a detailed assessment sheet (defined from the a priori visit to 10 dwellings) to collect information on building and dwelling characteristics. Participants will carry a smartphone with a GPS receiver and the Eco Emo tracker application permitting to identify their trips and visited places and to collect additional information on these trips (including their access to air conditioned). GPS data will permit to dynamically assess exposures in participants' everyday mobility. To move beyond simplistic assessments of personal heat stress, we will assess it in an ambulatory way considering personal ambient temperature, humidity, wind speed, and radiant temperature combined into the universal thermal climate index. Additionally, a meteorological station will be placed in the bedroom, while sensors measuring solar flux will be installed outdoor on the windows and balcony. Participants will also carry two bracelets for the measurement of physiological parameters (blood pressure, skin temperature, galvanic skin response as a marker of sweating, and heart rate). As part of the VF++ project, core temperature data will be additionally collected in a subsample of participants (e.g., 20 participants). Personal thermal discomfort, well-being, and sleep quality will be self-reported on the smartphone using the Eco Emo tracker application. An a posteriori phone questionnaire will collect detailed information on heat-related practices and health impacts over the observation period. Analyses of short-term effects will use repeated measure models. Investigations of momentary objective heat stress as the outcome will use statistical techniques for complex mixtures to handle the wide set of exposures. Analyses of sleep quality, well-being, and physiological measures as the outcomes will use two complementary designs: fixed-effect analyses of matched observations in the warm and in the cooler periods for the same participants; and participant-level fixed-effect analyses of pooled observations in the warm period. H3Sensing brings together epidemiologists, urbanists, and climate scientists. As research-to-policy translation, experts in urbanism involved in the project will formulate concrete technical recommendations and will identify practical solutions (in a pedagogical document of synthesis) to help urban actors willing to integrate considerations related to urban heat islands in their urbanistic regulations, public policies, and urban planning projects.

ELIGIBILITY:
Inclusion Criteria:

* Person aged between 30-64 years
* Person living in the Ile-de-France

Exclusion Criteria:

* Person subject to a legal protection measure (safeguarding of justice, curatorship, guardianship)
* Person deprived of liberty by a judicial or administrative decision,
* Person with a major functional limitation affecting their spatial mobility
* Person unable to complete a questionnaire
* Known cardiovascular (other than hypertension) or cerebrovascular disease: personal history of myocardial infarction, rhythm disorders or stroke
* People wearing a pacemaker or other implanted device, due to the risk of interference
* Pregnant or breastfeeding woman
* Person working night or shift
* Person with a definite plan to move in the coming months (before the second collection during summer)
* Person who initially refuses to participate in this second wave of the study
* Person working outside the Ile de France

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is a sample recruited through internet advertisement, residing in the Grand Paris, in warmer or cooler areas and in different types of dwellings.
  Quota sampling is applied in this research.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2035-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure | Measurement over 4 days, in two separate waves of 4 days
  Ambulatory blood pressure measured with a bracelet
Skin temperature | Measurement over 4 days, in two separate waves of 4 days
  It is measured with a bracelet, in degrees. It provides important information on the interaction of the body with the heat environment.
Accelerometry outcomes: total sleep time, sleep efficiency, and wake after sleep onset | These outcomes are collected for 5 successive nights in each of the two periods.
  These three accelerometry outcomes will be derived from a bracelet. Total sleep time is in hours and minutes. Sleep efficiency is a percentage. Wake after sleep onset is in minutes.

SECONDARY OUTCOMES:
Personal heat stress measured with the Universal Thermal Climate Index | Measured continuously over 2 waves of 4 days
  This secondary outcome will be measured with a unique indicator called the Universal Thermal Climate Index. Although it is based on 4 parameters measured with wearable sensors (air temperature, humidity, radiant temperature, and air flow), it is measured in degree Celsius (so with a unique unit).

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Louis Institute of Epidemiology and Public Health, Paris, France